CLINICAL TRIAL: NCT04403295
Title: Collaborative Specialty Care for Gulf War Illness
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 19-469
Record Dates: First submitted 2020-05-20; First posted 2020-05-27 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Gulf War Illness
Keywords: Veteran; Gulf War Illness; implementation; Chronic Pain; health coaching; problem-solving
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: In collaborative specialty care the specialty provider team will deliver health coaching and problem-solving treatment to GWVs and recommend the primary care team make monthly optimization of analgesics
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study coordinator conducting the randomization and study providers will not be blinded. Other staff and investigators (including the Principal Investigator) will be blind to study assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- collaborative specialty care (Experimental): In specialty collaborative care, the specialty provider team will deliver health coaching and problem-solving treatment to GWVs and recommend the primary care team make monthly optimization of analgesics.
  Interventions: Behavioral: Collaborative Specialty Care
- e-consultation (Active Comparator): In e-consultation the specialty provider team will make a onetime recommendation to the primary care team that the GWV locally receive health coaching and problem-solving treatment and analgesic optimization.
  Interventions: Behavioral: e-consultation

INTERVENTIONS:
Behavioral: Collaborative Specialty Care — In specialty collaborative care, the specialty provider team will deliver health coaching and problem-solving treatment to GWVs and recommend the primary care team make monthly optimization of analgesics.
  Arms: collaborative specialty care
Behavioral: e-consultation — In e-consultation the specialty provider team will make a onetime recommendation to the primary care team that the GWV locally receive health coaching and problem-solving treatment and analgesic optimization.
  Arms: e-consultation

SUMMARY:
Gulf War Veterans (GWVs) with Gulf War Illness (GWI) do not receive the care they should in the Veterans Affairs (VA). The investigators' data show 70% of GWVs with Gulf War Illness (GWI) do not receive treatment recommendations for their GWI and 78% are NOT very satisfied with their care. The quality of care GWVs receive must improve. VA and DoD have invested hundreds of millions of dollars to develop new treatments for GWVs, without effective delivery methods GWVs will not benefit. This study will be the first study to examine the best model of care to deliver treatments to GWVs with GWI. Determining the best model of care to translate research into practice is a key goal of the VA Gulf War Strategic Plan and a specific aim of this Request for Applications.

DETAILED DESCRIPTION:
There is a quality chasm between the care Gulf War Veterans (GWVs) should receive and the care they do receive. The investigators' data show 70% of GWVs with Gulf War Illness (GWI) do not receive treatment recommendations for their GWI and 78% are NOT very satisfied with their care. Reducing this quality chasm is essential. The VA and DoD have invested hundreds of millions of dollars to develop new treatments, including the second largest clinical trial for GWVs which is finding health coaching and problem-solving treatment both reduce the disability of GWI. Without effective models of healthcare to implement these treatments, GWVs will not benefit. In the current model of care, GWVs receive care locally through VA's primary care patient aligned care teams (PACTs). The VA War Related Illness and Injury Study Center (WRIISC) supports the current model of care by increasing local knowledge of the skills and treatments needed to manage GWI through national education efforts and electronic consultation (e-consultation) on difficult cases. The WRIISC and other stakeholders are currently questioning whether improving local knowledge of skills and treatments for GWI is enough to address the quality chasm, or if GWI is too complex to be treated in primary care without additional support from specialists in GWI. A potentially useful model of care for GWI is collaborative specialty care where specialists work with PACTs to synergistically treat patients. The local PACT is the lead of the team with the specialist providing some direct care to the patient (through tele-health) and also consulting with the PACT about other aspects of care. Collaborative specialty care is effective for other complex conditions (e.g., depression) with over 40 studies documenting its efficacy. The goal of this proposal is to conduct a hybrid type 1 randomized effectiveness/implementation trial for GWVs with GWI (n=220). The primary aim is to determine the effectiveness of tele-CSC as compared to e-consultation. In tele-CSC, the investigators' specialty provider team will deliver health coaching and problem-solving treatment to GWVs and recommend the PACT make monthly optimization of analgesics. In e-consultation the specialty provider team will make a onetime recommendation to the PACT that the GWV locally receive health coaching and problem-solving treatment and analgesic optimization. The secondary aim is to understand implementation outcomes. This information will be used to guide a future randomized (by VISN) multi-site implementation study. Throughout, an advisory committee of operations partners will be convened to ensure that the results of the study are able to directly and immediately improve care. Determining the best model of care to translate research into practice for GWVs with GWI is a key goal of the VA Gulf War Strategic Plan and a specific aim of this Request for Applications.

ELIGIBILITY:
Inclusion Criteria:

* deployed to Operation Desert Shield/Storm
* meets Kansas City (Steele) definition of GWI (which excludes conditions that may account for GWI)
* rates their activity limitations from pain at least 3 on a 0 to 10 point scale
* has a VA primary care provider

Exclusion Criteria:

* suicidal intent
* previous evaluation at the WRIISC or participated in our clinical trial for GWVs with GWI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Roland Morris Disability Scale | 6 months
  Pain disability will be assessed with the RMDS a 24 item scale of disability from pain. The RMDS is a core outcome measure for patients with chronic pain. A change of 2-3 points is considered clinically significant. Pain is present in 99% of GWVs with GWI and previous collaborative care trials in the VA have used this measure. Scores range from 0-24 with higher scores = greater disability.
World Health Organization Disability Schedule | 6 months
  The WHO-DAS 2.0 measures disability which is due to physical and mental health conditions. The WHO-DAS 2.0 is a 40 item measure that assesses 6 life tasks. The composite score will be used as the dependent variable. The items of the WHO-DAS have a factor loading on composite score of 0.82 to 0.98. The WHO-DAS was the primary outcome in our previous trial of problem-solving treatment and captures all over health disability. Scores range from 0-100 with higher scores equaling greater disability.

SECONDARY OUTCOMES:
Brief Pain Inventory - Interference Scale | 6 months
  The 7 item scale measures pain interference on mood, physical activity, social activity and other life activities. A one-point change is clinically significant. Scores range from 0-10 with higher scores equaling greater pain interference.
Patient Health Questionnaire Somatic Symptom Scale - 15 | 6 months
  The PHQ-15 captures somatic symptoms. The PHQ-15 was validated on a sample of 6,000 and found to be reliable, valid and responsive to change. Scores range from 0-30 and higher scores are greater symptom severity.
Patient Activation Measure | 6 months
  The PAM is a 13 item self-report measure of the patient's active engagement in self-management their health. The PAM is reliable and valid. Scores range from 0-100 with higher scores indicating greater activation.
Satisfaction: Patient Satisfaction Questionnaire | 6 month
  The PSQ-III is a 50-item self-report measure with 7 subscales reliability with ranges from .77-.89. The investigators will use the composite score. Score range from 0-100 with higher scores indicating greater satisfaction.
Roland Morris Disability Scale | 9 month
  Pain disability will be assessed with the RMDS a 24 item scale of disability from pain. The RMDS is a core outcome measure for patients with chronic pain. A change of 2-3 points is considered clinically significant. Pain is present in 99% of GWVs with GWI and previous collaborative care trials in the VA have used this measure. Scores range from 0-24 with higher scores = greater disability.
World Health Organization Disability Schedule | 9 month
  The WHO-DAS 2.0 measures disability which is due to physical and mental health conditions. The WHO-DAS 2.0 is a 40 item measure that assesses 6 life tasks. The composite score will be used as the dependent variable. The items of the WHO-DAS have a factor loading on composite score of 0.82 to 0.98. The WHO-DAS was the primary outcome in our previous trial of problem-solving treatment and captures all over health disability. Scores range from 0-100 with higher scores equaling greater disability.
Brief Pain Inventory - Interference Scale | 9 month
  The 7 item scale measures pain interference on mood, physical activity, social activity and other life activities. A one-point change is clinically significant. Scores range from 0-10 with higher scores equaling greater pain interference.
Patient Health Questionnaire Somatic Symptom Scale - 15 | 9 month
  The PHQ-15 captures somatic symptoms. The PHQ-15 was validated on a sample of 6,000 and found to be reliable, valid and responsive to change. Scores range from 0-30 and higher scores are greater symptom severity.
Patient Activation Measure | 9 month
  The PAM is a 13 item self-report measure of the patient's active engagement in self-management their health. The PAM is reliable and valid. Scores range from 0-100 with higher scores indicating greater activation.
Satisfaction: Patient Satisfaction Questionnaire | 9 month
  The PSQ-III is a 50-item self-report measure with 7 subscales reliability with ranges from .77-.89. The investigators will use the composite score. Score range from 0-100 with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Marie McAndrew, PhD, Principal Investigator — East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ; Justeen K Hyde, PhD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA; Scott E. Sherman, MD MPH, Principal Investigator — VA NY Harbor Healthcare System, New York, NY
Locations (1):
- East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ, East Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schneider AH, Bair MJ, Helmer DA, Hyde J, Litke D, Lu SE, Rogers ES, Sherman SE, Sotolongo A, Anastasides N, Sullivan N, Graff F, McAndrew LM. Protocol for a type 1 hybrid effectiveness/implementation clinical trial of collaborative specialty care for Veterans with Gulf War Illness. Life Sci. 2022 Mar 1;292:120004. doi: 10.1016/j.lfs.2021.120004. Epub 2021 Sep 29. PMID 34599935
- [Result] Lesnewich LM, Hyde JK, McFarlin ML, Bolton RE, Bayley PJ, Chandler HK, Helmer DA, Phillips LA, Reinhard MJ, Santos SL, Stewart RS, McAndrew LM. 'She thought the same way I that I thought:' a qualitative study of patient-provider concordance among Gulf War Veterans with Gulf War Illness. Psychol Health. 2025 Apr;40(4):616-634. doi: 10.1080/08870446.2023.2248481. Epub 2023 Sep 1. PMID 37654203

DOCUMENTS (1):
  • Informed Consent Form (2024-05-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT04403295/ICF_000.pdf